CLINICAL TRIAL: NCT02649725
Title: Prospective Questionnaire Based Observational Study Measuring the Degree of Patient's Satisfaction With the Outcomes of Expensive Cytotoxic Agents.
Brief Title: Patients Satisfaction With the Outcomes of Expensive Cytotoxic Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: International Medical Center of Egypt. (Unknown); Metghamr Cancer Center. (Unknown); Benha University (Other); Misr University for Science and Technology (Other); Kuwait Cancer Control Center (Other)
Responsible Party: Principal Investigator, Mahmoud Ellithy, Associate professor of clinical oncology.Faculty of Medicine., Ain Shams University
Other Study IDs: Cure and more2
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Patient's Satisfaction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: patient's satisfaction — Questionnaire based measurement.

SUMMARY:
The purpose of this study is to determine whether there is positive (beneficial) impact of expensive cytotoxic agents on the cancer patients. It is a questionnaire based study that will be filled by the cancer patients without obligations.

DETAILED DESCRIPTION:
This is a prospective observational questionnaire based study measuring the degree of patient satisfaction with the outcomes of some expensive cytotoxic agents.

The tested drugs are trastuzumab, lapatinib, sunitinib, m tor inhibitors, sorafenib, cetuximab, panitumumab, bevacizumab, erlotinib, rituximab, imatinib mesylate, gefitinib, abiraterone acetate, cabazitaxel, pertuzumab, fulvestrant, pemetrexate and crizotinib.

The evaluation will be through a predesigned template questionnaire that will be applied to all the tested drugs. The questions are divided into five categories measuring five items, the negative impact of the drug on patient's finances, satisfaction with drug efficacy, toxicity and effect on quality of life, satisfaction with drug availability in the market and satisfaction with the received education from the treating physician about the drug before usage. A predesigned questionnaire based scoring system will categorizes the processed data to low, intermediate and high score for each of the five measured topics. The data will be processed and each drug will acquire low, moderate or high score. Subsequent recommendations for revision of the drug price, cost effective analysis studies, physician education about drug pharmaceutical perspectives will be elaborated for some drugs. The study will clarify the most annoying and frequently reported side effect for each drug and will suggest recommendations for its treatment.

The study is currently recruiting patients.

The study is currently accepting to add authors (Oncology physicians) who can fulfill the following prerequisites:

1. Answer a questionnaire that will be mailed to him upon request and propagate this questionnaire to 10 oncology physicians in his center to answer them. (The 11 questionnaires should be scanned and mailed to ellithym@med.asu.edu.eg. or given as hard copies to Dr Mahmoud Ellithy (Mobile: +01000069694).

   (This questionnaire is designed to be answered by oncology physicians to measure their degree of satisfaction with the outcomes of expensive cytotoxic agents).

   The questionnaire can be answered electronically online https://www.surveymonkey.com/r/Cureandmore. (for oncologist with foreign nationality who want to share as an author. Egyptian oncologists should fill a hard copy not online).

   Disclosure: The Questionnaire for the physicians is a clinical trial registered clinical trials.gov with NCT02630979. URL. https://clinicaltrials.gov/ct2/show/nct02630979.
2. Each author must share with at least 90 patients with at least 5 patients for each drug. The maximum allowed numbers of authors from each center are two authors sharing with 180 patients till closure of the study in 30th January 2019.
3. Share with any new idea that will add benefit to the study. ( Item 1 and 2 are mandatory).

The Oncologist who want to share as an author in this study must sign a memorandum of aggrement consenting for the accuracy, confidentiality and validity of the data with a copyright, stating that he must obtain a written permission from the research team (Cure and More research team) to produce any text, figures, tables or illustrations from this study in future works of his own.

ELIGIBILITY:
Inclusion criteria:

1. The patient should be willing to share in the study.
2. The patient should have full mental power to answer the questionnaire.
3. Adult from 17 to 70 years.
4. Patient should be able to complete the course of treatment without interruption due to financial issues or other issues like transportation obstacles.

Exclusion criteria:

1. The patient with psychological disease that impairs credibility of his answer.
2. Patient with special requirements/difficulties with communications.
3. Patient who have difficulty with their memory e.g. recall of events, learning new things, remembering appointments.
4. Patient who have epilepsy blackouts or dizzy spills.
5. Patient who have any visual impairment other than standard glasses.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients who are willing to answer the questionnaire voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The patient's satisfaction questionnaire | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Elbaghdady, Specialis, Study Director — Misr University for Science and Technology
Locations (1):
- Faculty of Medicine. AIn Shams University, Cairo, Elabbasia, Egypt

IPD SHARING:
Plan to Share IPD: No